CLINICAL TRIAL: NCT00448019
Title: Fludarabine, Cyclophosphamide, Rituximab and Bevacizumab in the Treatment of Relapsed Chronic Lymphocytic Leukemia
Brief Title: FCR and Bevacizumab in the Treatment of Relapsed Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDACC-2005-0992; NCI-2010-00591 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Fludarabine; Cyclophosphamide; Rituximab; Bevacizumab; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Rituximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCR + Bevacizumab (Experimental): FCR = Fludarabine 25 mg/m^2 intravenous (IV) , Cyclophosphamide 250 mg/m^2 IV daily for 3 days, Rituximab 375 mg/m^2 IV Day 1, followed by 500 mg/m^2 IV. FCR daily for 3 days. Bevacizumab 10 mg/Kg IV on Day 3, course 1.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 IV over 30 minutes daily for 3 days
  Other Names: Fludara; Fludarabine Phosphate
Drug: Cyclophosphamide — 250 mg/m^2 IV over 30 minutes daily for 3 days
  Other Names: Cytoxan; Neosar
Drug: Rituximab — 375 mg/m^2 IV on Day 1 by prolonged infusion. All subsequent doses 500 mg/m^2 IV 30-minute infusion.
  Other Names: Rituxan
Drug: Bevacizumab — 10 mg/Kg IV on Day 3, course 1 over 30-90 minutes
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF

SUMMARY:
The goal of this clinical research study is to learn if the combination of fludarabine, cyclophosphamide, rituximab, and bevacizumab is effective in treating chronic lymphocytic leukemia in patients who have already been treated with chemotherapy. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
During the study, you will have up to 6 "cycles" of treatment. A cycle is made up of treatment with the study drugs for 3-4 days and then about 3-1/2 weeks (25 days) of no treatment (about 4 weeks total). Treatment with the study drugs will be given for 4 days in a row on the first cycle, and 3 days in a row on Cycles 2-6. On Day 1 of each cycle, you will receive rituximab through a needle in a vein. On Cycle 1, since it is your first exposure to rituximab, it must be given slowly, so it may take 6-8 hours to complete. On the cycles after that, it can be given more rapidly, over 3-4 hours. Cyclophosphamide and fludarabine will be given separately through a needle in a vein on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2-6. Cyclophosphamide and fludarabine will each be given over 30 minutes. Bevacizumab will be given through a needle in a vein over 90 minutes on Day 3 of Cycle 1. If it is well tolerated, the next dose of Bevacizumab will be given over 60 minutes on Day 2 of Cycle 2. If the Cycle 2 dose is well tolerated, the next doses of Bevacizumab will be given over 30 minutes on Day 2 of Cycles 2-6. In addition to the study drugs, you may also be given fluids by vein to help flush the kidneys, to help prevent possible kidney damage. You may receive up to 6 cycles of treatment. Treatment will be given on an outpatient basis. The injections for each daily treatment visit should take less than 6 hours.

Up to 66 patients will take part in the study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell CLL
* Relapsed, fludarabine-sensitive (duration of response > 6 months as assessed by prior treating physician) or fludarabine-naive patients
* Rai Stage III or IV, or Rai Stage I or II if determined to have disease progression as evidenced by rapid doubling of peripheral lymphocyte count, progressive lymphadenopathy, progressive splenomegaly, or B symptoms.
* Prestudy WHO Performance Status </= 2.
* Signed, written Institutional Review Board (IRB)approved informed consent.
* Men and women of reproductive potential must agree to follow accepted birth control methods during treatment and for 3 months after completion of treatment.
* Acceptable liver function: Bilirubin </= 2.0 mg/dL (26 umol/L), AST (SGOT) and/or ALT (SGPT) </= 2 times upper limit of normal.
* Acceptable hematologic status: Platelet count >/= 50 x 10^9/L., absolute neutrophil count (ANC) >/= 1 x 10^9/L.
* Acceptable renal function: Serum creatinine </= 2.0 mg/dL

Exclusion Criteria:

* Cancer radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or other investigational therapy within 4 weeks prior to Study Day 1.
* Known infection with HIV, hepatitis B, or hepatitis C
* Transformation to aggressive B-cell malignancy (e.g., large B-cell lymphoma, Richter's Syndrome, or prolymphocyte leukemia [PLL]).
* Patients with secondary malignancy requiring active treatment (except hormonal therapy).
* Active uncontrolled bacterial, viral, or fungal infections.
* New York Heart Association Class II-IV cardiac disease or myocardial infarction within the past 6 months prior to Study Day 1.
* Pregnant or currently breast-feeding.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study.
* Blood pressure of > 150/100 mmHg
* Unstable angina
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 1.
* Urine protein:creatinine ratio >/= 1.0 at screening.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1.
* Serious, non-healing wound, ulcer, or bone fracture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan O'Brien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Jain P, Lee HJ, Qiao W, Wierda W, Benjamini O, Burger J, Ferrajoli A, Estrov Z, Kantarjian H, Keating M, O'Brien S. FCR and bevacizumab treatment in patients with relapsed chronic lymphocytic leukemia. Cancer. 2014 Nov 15;120(22):3494-501. doi: 10.1002/cncr.28910. Epub 2014 Jul 15. PMID 25043749
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 23, 2007 to November 17, 2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | FCR + Bevacizumab
Started | 64
Completed | 57
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Disease progression | 1
Not completed — Death | 2
Not completed — Insurance Issues | 1

BASELINE CHARACTERISTICS:
Population: Two participants included in the study demographics were registered but withdrew prior to receiving treatment.
Arm/Group | FCR + Bevacizumab
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate
Description: Progression free survival (PFS) was defined as the time from the start of treatment to progression, which included treatment failure, relapse, or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Baseline up to 5 years
Population: Five participants of the 62 treated participants were not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | FCR + Bevacizumab
Number analyzed (Participants) | 57
Months | 13.5 [1 to 50]

2. Secondary Outcome: Number of Participants With Complete or Partial Response to Fludarabine, Cyclophosphamide, Rituximab, and Bevacizumab Therapy in Previously Treated Chronic Lymphocytic Leukemia (CLL)
Description: Response criteria for Complete response (CR) - Nodes: None; Liver/Spleen Size: Not palpable; Symptoms: None; polymorphonuclear leukocytes (PMN): >1,500/μl; Platelets >100,000/μl; Hemoglobin (untransfused): >11,0 g/dl; Lymphocytes: <4,000/μl; Bone Marrow aspirate: <30% lymphocytes; Biopsy: No lymphocyte infiltrate; and for Partial Response (PR), Nodes: >/= 50% decrease; Liver/Spleen Size: >/= 50% decrease; Symptoms: None; Platelets >100,000/μl or > 50% improvement from baseline; Hemoglobin (untransfused): >11.0 g/dl or >50% improvement from baseline; Lymphocytes: >50% decrease; Biopsy: <30% lymphocytes with residual disease on biopsy for nodular PR (NPR).
Time Frame: Response assessed after three 4-week courses and after six courses, up to 24 weeks
Population: Five participants of the 62 treated participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | FCR + Bevacizumab
Number analyzed (Participants) | 57
participants
  Complete Response (CR) | 13
  Partial Response (PR) | 24
  Nodular Partial Response (NPR) | 8

3. Secondary Outcome: Overall Response Rate (ORR) to Fludarabine, Cyclophosphamide, Rituximab, and Bevacizumab Therapy in Previously Treated CLL
Description: ORR defined as CR and PR response where response criteria for Complete response (CR) - Nodes: None; Liver/Spleen Size: Not palpable; Symptoms: None; polymorphonuclear leukocytes (PMN): >1,500/μl; Platelets >100,000/μl; Hemoglobin (untransfused): >11,0 g/dl; Lymphocytes: <4,000/μl; Bone Marrow aspirate: <30% lymphocytes; Biopsy: No lymphocyte infiltrate; and for Partial Response (PR), Nodes: >/= 50% decrease; Liver/Spleen Size: >/= 50% decrease; Symptoms: None; Platelets >100,000/μl or > 50% improvement from baseline; Hemoglobin (untransfused): >11.0 g/dl or >50% improvement from baseline; Lymphocytes: >50% decrease; Biopsy: <30% lymphocytes with residual disease on biopsy for nodular PR (NPR).
Time Frame: Response assessed after three 4-week courses and after six courses, up to 24 weeks
Population: Five participants of the 62 treated participants were not evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | FCR + Bevacizumab
Number analyzed (Participants) | 57
percentage of participants | 79

ADVERSE EVENTS:
Time Frame: Participants evaluated for adverse events at each study visit for study duration, up to six courses of 4 weeks. Overall collection period: May 2011 to September 2014.
Arm/Group | FCR + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 33/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FCR + Bevacizumab (N=62)
Anemia (Blood and lymphatic system disorders) | 1
Gastrointestinal hemorrhage (Blood and lymphatic system disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 4
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Pain (General disorders) | 1
Tumor lysis Syndrome (General disorders) | 1
Herpes simplex II (Infections and infestations) | 1
Infection (Infections and infestations) | 3
Neutropenic Fever (Infections and infestations) | 10
pneumonia (Infections and infestations) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FCR + Bevacizumab (N=62)
Neutropenia (Blood and lymphatic system disorders) | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Infection (Infections and infestations) | 30
Nausea and vomiting (Gastrointestinal disorders) | 22
Fatigue (General disorders) | 16
Anemia (Blood and lymphatic system disorders) | 9
Gastrointestinal Hemorrhage (Blood and lymphatic system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Blurred vision (Eye disorders) | 2
Syncope (Nervous system disorders) | 1
Hypertension (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less